CLINICAL TRIAL: NCT02354404
Title: Phase 1B, Open-Label, Clinical Trial to Evaluate Safety, Tolerability and Immunogenicity of the Investigational Ebola Vaccines, VRC-EBOADC069-00-VP, VRC-EBOADC076-00-VP and VRC-EBOMVA079-00-VP in Healthy Adults in Kampala Uganda
Brief Title: Clinical Trial of Ebola Vaccines cAd3-EBO, cAd3-EBOZ and MVA-EbolaZ in Healthy Adults in Uganda
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: US Military HIV Research Program (Network); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RV 422
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-09

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Ebola virus; Filoviridae Infections; Hemorrhagic Fever, Ebola; Viral Diseases; Hemorrhagic Fevers, Viral
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Filoviridae Infections; Virus Diseases; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1a: cAd3-EBOZ at 1x10(10) PU (Experimental): Part 1: cAd3-EBOZ at 1x10(10) PU intramuscularly at Day 0; Part 2: Option to receive MVA-EbolaZ at 1x10(8) PFU intramuscularly after Study Week 36 as a boost to the Part 1 study vaccination
  Interventions: Biological: cAd3-EBOZ; Biological: MVA-EbolaZ
- Group 1b: cAd3-EBOZ at 1x10(11) PU (Experimental): Part 1: cAd3-EBOZ at 1x10(11) PU intramuscularly at Day 0; Part 2: Option to receive MVA-EbolaZ at 1x10(8) PFU intramuscularly after Study Week 36 as a boost to the Part 1 study vaccination
  Interventions: Biological: cAd3-EBOZ; Biological: MVA-EbolaZ
- Group 1c: cAd3-EBO at 2x10(10) PU (Experimental): Part 1: cAd3-EBO at 2x10(10) PU intramuscularly at Day 0; Part 2: Option to receive MVA-EbolaZ at 1x10(8) PFU intramuscularly after Study Week 36 as a boost to the Part 1 study vaccination
  Interventions: Biological: cAd3-EBO; Biological: MVA-EbolaZ
- Group 1d: cAd3-EBO at 2x10(11) PU (Experimental): Part 1: cAd3-EBO at 2x10(11) PU intramuscularly at Day 0; Part 2: Option to receive MVA-EbolaZ at 1x10(8) PFU intramuscularly after Study Week 36 as a boost to the Part 1 study vaccination
  Interventions: Biological: cAd3-EBO; Biological: MVA-EbolaZ
- Group 2a:cAd3-EBO at 2x10(10) PU (Experimental): Part 1: cAd3-EBO at 2x10(10) PU intramuscularly at Day 0 (as a boost to prior receipt of the Ebola DNA WT vaccine); Part 2: Option to receive MVA-EbolaZ at 1x10(8) PFU intramuscularly after Study Week 36 as a boost to the Part 1 study vaccination
  Interventions: Biological: cAd3-EBO; Biological: MVA-EbolaZ
- Group 2b: cAd3-EBO at 2x10(11) PU (Experimental): Part 1: cAd3-EBO at 2x10(11) PU intramuscularly at Day 0 (as a boost to prior receipt of the Ebola DNA WT vaccine); Part 2: Option to receive MVA-EbolaZ at 1x10(8) PFU intramuscularly after Study Week 36 as a boost to the Part 1 study vaccination
  Interventions: Biological: cAd3-EBO; Biological: MVA-EbolaZ

INTERVENTIONS:
Biological: cAd3-EBOZ — cAd3 vaccine vector expressing Ebola glycoprotein from the Zaire strain in single dose vials at 1x10(11) PU/mL.
  Other Names: VRC-EBOADC076-00-VP
  Arms: Group 1a: cAd3-EBOZ at 1x10(10) PU; Group 1b: cAd3-EBOZ at 1x10(11) PU
Biological: cAd3-EBO — 1:1 ratio of cAd3 vaccine vectors expressing Ebola glycoprotein from the Zaire and Sudan strains filled into single dose vials at 1x10(11) PU/mL of each [2x10(11) PU/mL total].
  Other Names: VRC-EBOADC069-00-VP
  Arms: Group 1c: cAd3-EBO at 2x10(10) PU; Group 1d: cAd3-EBO at 2x10(11) PU; Group 2a:cAd3-EBO at 2x10(10) PU; Group 2b: cAd3-EBO at 2x10(11) PU
Biological: MVA-EbolaZ — MVA vaccine vector that expresses Ebola glycoprotein from the Zaire strain in single dose vials at 3.2 x 10(8) PFU/mL
  Other Names: VRC-EBOMVA079-00-VP

SUMMARY:
Phase Ib study in 90 healthy adults,18 years to 65 years of age, to evaluate the safety, tolerability and immunogenicity of the VRC-EBOADC069-00-VP (cAd3-EBO) and VRC-EBOADC076-00-VP (cAd3-EBOZ) investigational Ebola vaccines in Part 1 and boosting with the VRC-EBOMVA079-00-VP (MVA-EbolaZ) investigational Ebola vaccine in Part 2.

Part 1: Randomizations to cAd3-EBO or cAd3-EBOZ at two different dose levels within Group 1 will include at least 60 volunteers who have never received an investigational Ebola vaccine. Randomizations to cAd3-EBO at two different dose levels within Group 2 may include up to 30 eligible participants who previously participated in the RV247 vaccine clinical trial and received the investigational VRC-EBODNA023-00-VP (Ebola DNA WT) vaccine.

Part 2: Participants in Part 1 may receive a booster vaccination with the MVA-EbolaZ vaccine at the same dose level.

DETAILED DESCRIPTION:
Study Design: This Phase 1b, open-label study to examine safety, tolerability and immunogenicity of investigational Ebola vaccines is conducted in two Parts. In Part 1 subjects are randomized to receive either the cAd3-EBO or cAd3-EBOZ vaccine at two different dose levels. In Part 2, participants from Part 1 may receive a booster injection with the MVA-EbolaZ vaccine; all at the same dose level. The hypotheses are that the study vaccines, cAd3-EBO, cAd3-EBOZ and MVA-EbolaZ, will be safe and will elicit immune responses to Ebola glycoprotein (GP). The primary objectives are to evaluate the safety and tolerability of the study vaccines administered as intramuscular (IM) injections. The secondary objectives are related to immunogenicity.

Study Products Description:

VRC-EBOADC069-00-VP (cAd3-EBO) is composed of two recombinant cAd3 vectors in a 1:1 ratio that express Ebola WT GPs from Zaire and Sudan strains. It is formulated at 2x10(11) particle units (PU)/mL.

VRC-EBOADC076-00-VP (cAd3-EBOZ) is composed of a cAd3 vector that expresses Ebola WT GP from the Zaire strain. It is formulated at 1x10(11) PU/mL.

VRC-DILADC065-00-VP (diluent) is the vaccine formulation buffer and will be used when needed to prepare the correct dosage of cAd3-EBO or cAd3-EBOZ.

VRC-EBOMVA079-00-VP (MVA-EbolaZ) is composed of a MVA vector that expresses Ebola WT GP from the Zaire strain. It is formulated at 3.2x10(8) PFU/mL.

Part 1 Study Plan:

Group 1: 60 volunteers will be randomized: 15 in each of the two dosage groups for VRC-EBOADC069-00-VP [2x10(10) PU or 2x10(11) PU] and 15 in each of the two dosage groups for VRC-EBOADC076-00-VP [1x10(10) PU or 1x10(11) PU].

Group 2: up to 30 volunteers that previously participated in the RV 247 clinical trial who received the investigational product VRC-EBODNA023-00-VP will be randomized to receive one of the two dosage groups for VRC-EBOADC069-00-VP.

The two groups will be enrolled simultaneously. If less then 30 participants enroll into Group 2, additional participants may be enrolled into Group 1 for a total of 90 participants overall. Participants will be evaluated by 9 clinic visits over 48 weeks.

Part 2 Study Plan:

Part 1 participants who received a study vaccination and have completed at least 36 weeks of follow-up, who are eligible and consent may receive a booster injection with the VRC-EBOMVA079-00-VP vaccine at 1x10(8) particle forming units (PFU). Participants will be evaluated by 11 clinic visits over 48 weeks after beginning Part 2.

ELIGIBILITY:
Part 1 Inclusion Criteria:

A volunteer subject must meet all of the following criteria:

* 18 to 65 years old.
* Available for clinical follow-up through Week 48.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* Must be willing to be taken home at enrollment visit and allow home visits if participant does not keep appointments
* Must complete an Assessment of Understanding successfully.
* Able to read (English or Luganda) and willing to complete the informed consent process.
* Willing to donate blood for sample storage to be used for future research.
* In good general health without clinically significant medical history.
* Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) ≤ 40 within the 56 days prior to enrollment.

Laboratory Inclusion Criteria within 56 days prior to enrollment:

* Hemoglobin ≥ 11.0 g/dL for women; ≥12.5 g/dL for men.
* White blood cells (WBC) = 2,500-12,000 cells/mm3.
* WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
* Total lymphocyte count ≥ 800 cells/mm3.
* Platelets = 125,000 - 400,000/mm3.
* Alanine aminotransferase (ALT) ≤ 1.25 x upper limit of normal (ULN).
* Serum creatinine ≤ 1 x ULN.
* Partial thromboplastin time (PTT) within institutional normal range.
* Prothrombin time (PT) within institutional normal range.
* HIV-uninfected as evidenced by a negative FDA-approved HIV diagnostic test.

Female-Specific Inclusion Criteria:

* Negative β-HCG (human chorionic gonadotropin) pregnancy test on day of enrollment.
* Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 24 weeks after study vaccination if presumed to be of reproductive potential.

Part 1 Exclusion Criteria:

Volunteer has received any of the following substances:

* Investigational Ebola or Marburg vaccine (other than the Ebola DNA vaccine delivered in RV 247) in a prior clinical trial or prior receipt of a cAd3 adenoviral vectored investigational vaccine.
* Chronic use of immunomodulators and systemic glucocorticoids in daily doses of glucocorticoid equivalence > 20 mg of prednisolone, for periods exceeding 10 days. Non-steroidal anti-inflammatory drugs [NSAIDS] are permitted.
* Participants that have used less than the stated glucocorticoid dose may still be excluded at the Investigator's discretion.
* Blood products within 112 days prior to enrollment.
* Investigational research agents within 28 days prior to enrollment.
* Live attenuated vaccines within 28 days prior to enrollment.
* Subunit or killed vaccines within 14 days prior to enrollment.
* Current anti-tuberculosis prophylaxis or therapy.

Female-Specific Exclusion Criteria:

* Woman who is breast-feeding or planning to become pregnant during the first 24 weeks after study vaccine administration.

Volunteer has a history of any of the following clinically significant conditions:

* Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
* Clinically significant autoimmune disease or immunodeficiency.
* Asthma that is not well controlled.
* Diabetes mellitus (type I or II), with the exception of gestational diabetes.
* Thyroid disease that is not well controlled.
* A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
* Idiopathic urticaria within the last 1 year.
* Hypertension that is not well controlled.
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
* Malignancy that is active or history of a malignancy that is likely to recur during the period of the study.
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years.
* Asplenia or functional asplenia.
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within five years prior to enrollment, history of a suicide plan or attempt.
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Part 2 Inclusion Criteria:

* Received the Part 1 study injection and is willing to participate in Part 2.
* Satisfactory completion of the Assessment of Understanding
* Subject is assessed by the Site Principal Investigator or designee as in good general health without clinically significant medical history that precludes participation.

Female-Specific Inclusion Criteria:

* Negative β-HCG pregnancy test on day of enrollment if presumed to be of reproductive potential.
* Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 24 weeks after study vaccination if presumed to be of reproductive potential.

Part 2 Exclusion Criteria:

* Type 1 hypersensitivity to aminoglycosides antibiotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events after vaccination | 7 days
  Incidence is reported for solicited events for 7 days after each vaccination.
Incidence of unsolicited adverse events of any severity 28 days after vaccination | 28 days
  Incidence is reported for unsolicited events for 28 days after each vaccination. The reporting period is Day 0 to Day 28.
Incidence of serious adverse events or new chronic medical conditions through the last study visit | From first study injection through 48 weeks after final study injection
  Incidence is reported of serious adverse events and new chronic medical conditions for 48 weeks after vaccination.
Mean change from baseline in safety laboratory measures | 28 days after each vaccination
  At Days 2 or 3, 14, and 28 blood will be drawn to measure safety measures that many include complete blood count (CBC), creatinine, ALT, PT and PTT.

SECONDARY OUTCOMES:
Antibody response to Ebola GP as measured by ELISA | 4 weeks after each vaccination
  Blood is collected at baseline and 4 weeks after vaccination
Antibody response to Ebola GP as measured by neutralization assay | 4 weeks after vaccination
  Blood is collected at baseline and 4 weeks after vaccination
T cell immune response measured by intracellular cytokine staining (ICS) | 4 weeks after vaccination
  Blood is collected at baseline and 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Merlin Robb, MD, Study Chair — US Military HIV Research Program; Julie Ledgerwood, DO, Study Chair — VRC, NIAID, NIH
Locations (1):
- Makerere University Walter Reed Project, Kampala, Uganda

REFERENCES:
- [Background] Kibuuka H, Berkowitz NM, Millard M, Enama ME, Tindikahwa A, Sekiziyivu AB, Costner P, Sitar S, Glover D, Hu Z, Joshi G, Stanley D, Kunchai M, Eller LA, Bailer RT, Koup RA, Nabel GJ, Mascola JR, Sullivan NJ, Graham BS, Roederer M, Michael NL, Robb ML, Ledgerwood JE; RV 247 Study Team. Safety and immunogenicity of Ebola virus and Marburg virus glycoprotein DNA vaccines assessed separately and concomitantly in healthy Ugandan adults: a phase 1b, randomised, double-blind, placebo-controlled clinical trial. Lancet. 2015 Apr 18;385(9977):1545-54. doi: 10.1016/S0140-6736(14)62385-0. Epub 2014 Dec 23. PMID 25540891
- [Background] Ledgerwood JE, DeZure AD, Stanley DA, Coates EE, Novik L, Enama ME, Berkowitz NM, Hu Z, Joshi G, Ploquin A, Sitar S, Gordon IJ, Plummer SA, Holman LA, Hendel CS, Yamshchikov G, Roman F, Nicosia A, Colloca S, Cortese R, Bailer RT, Schwartz RM, Roederer M, Mascola JR, Koup RA, Sullivan NJ, Graham BS; VRC 207 Study Team. Chimpanzee Adenovirus Vector Ebola Vaccine. N Engl J Med. 2017 Mar 9;376(10):928-938. doi: 10.1056/NEJMoa1410863. Epub 2014 Nov 26. PMID 25426834
- [Background] Sarwar UN, Costner P, Enama ME, Berkowitz N, Hu Z, Hendel CS, Sitar S, Plummer S, Mulangu S, Bailer RT, Koup RA, Mascola JR, Nabel GJ, Sullivan NJ, Graham BS, Ledgerwood JE; VRC 206 Study Team. Safety and immunogenicity of DNA vaccines encoding Ebolavirus and Marburgvirus wild-type glycoproteins in a phase I clinical trial. J Infect Dis. 2015 Feb 15;211(4):549-57. doi: 10.1093/infdis/jiu511. Epub 2014 Sep 14. PMID 25225676